CLINICAL TRIAL: NCT04635696
Title: Evaluating the Efficacy of Ethyl Chloride on Patients' Reported Pain With Negative Pressure Wound Therapy
Brief Title: Ethyl Chloride for NPWT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ProMedica Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-079
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Ethyl Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethyl Chloride (Experimental): Ethyl Chloride topical anesthetic mist will be sprayed on the area of adhesive during dressing change for patients with negative pressure wound therapy
  Interventions: Drug: Ethyl chloride
- Tissue culture grade water (Placebo Comparator): Tissue culture grade water (Nature's Tears Eyemist) will be sprayed on the area of adhesive during dressing change for patients with negative pressure wound therapy
  Interventions: Other: Tissue culture grade water

INTERVENTIONS:
Drug: Ethyl chloride — Pressurized vapocoolant developed for acute, mild pain relief.
  Other Names: vapocoolant
  Arms: Ethyl Chloride
Other: Tissue culture grade water — Pressurized water mist
  Other Names: Nature's Tears Eyemist
  Arms: Tissue culture grade water

SUMMARY:
Negative pressure wound therapy (NPWT) has been shown to improve wound care outcomes for acute and chronic wounds as well as for surgical incision sites. We have found that patients report significant pain during dressing changes specifically with the removal of the clear adhesive drape. Upon review of the literature, there were multiple studies related to pain and the removal of the sponge (filler) but limited studies relating to the pain associated with the removal of the drape. The patient reported pain with drape removal has led to increased psychological stress and decreased compliance with the dressing change protocol. Application of a topical anesthetic to the drape during the dressing change has the potential to decrease the pain experienced by the patient. An FDA approved ethyl chloride spray is a topical anesthetic that can be sprayed onto the outer perimeter of the drape during the dressing change as a means to decrease pain. We hypothesize that the use of ethyl chloride spray will result in patients experiencing less pain leading to decreased psychological stress, improved compliance with dressing changes, and overall improved customer satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* an orthopaedic/trauma wound and/or surgical incision
* treatment with NPWT as a hospital inpatient
* minimum of at least one NPWT dressing changes or discontinuation of NPWT prior to discharge.
* dressing change in enterostomal therapy department

Exclusion Criteria:

* cognitive impairment preventing informed consent
* history of hypersensitivity to cold/vapocoolant
* outpatient NPWT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Patient-reported post procedure pain | immediately after drape removal
  Pain reported on 0-10 numeric pain scale (NPS), where lower reported scores are favorable.
Patient-reported during procedure pain | during drape removal
  Pain reported on 1-10 numeric pain scale (NPS), where lower reported scores are favorable.

SECONDARY OUTCOMES:
Change in pain score from pre-procedure to post-procedure | immediately prior to drape change to immediately following drape change
  change in pain reported on 0-10 numeric pain scale (NPS), where lower reported scores are favorable.
Change in pain score from pre-procedure to during procedure | immediately prior to drape change to during drape change
  change in pain reported on 0-10 numeric pain scale (NPS), where lower reported scores are favorable.

CONTACTS AND LOCATIONS:
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tank JC, Georgiadis GM, Bair JM, Rice A, O'Mara Gardner K, Chen JT, Redfern RE. Does The Use of Ethyl Chloride Improve Patient-Reported Pain Scores With Negative Pressure Wound Therapy Dressing Changes? A Prospective, Randomized Controlled Trial. J Trauma Acute Care Surg. 2021 Jun 1;90(6):1061-1066. doi: 10.1097/TA.0000000000003157. PMID 33755640